CLINICAL TRIAL: NCT05111418
Title: Myocardial Bridge Evaluation Towards Personalised Medicine: the RIALTO Registry
Acronym: RIALTO
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, DAMARIO DOMENICO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3812
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Myocardial Bridge
Keywords: Myocardial Bridge; MACE; Ischemia; Beta-blockers; Coronary angiography; Personalised medicine
MeSH Terms: conditions — Myocardial Bridging; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myocardial bridge (MB) is a congenital anomaly of epicardial circulation characterized by an intramural course of a coronary segment. This anatomical arrangement causes the artery to be squeezed during systole potentially causing flow impairment and ischemia. For this study, MB is defined as the presence of systolic compression in an epicardial vessel causing at least 50% of caliber reduction from diastole. MB can be disabling as it worsens the quality of life. Early detection of this congenital condition is crucial, and an invasive functional assessment of the ischemic burden should be considered to evaluate the need for medical or surgical therapy.

This is an observational study, involving four Italian centres. Study Objectives are: To assess the risk of future cardiovascular complications in patients with MB referred for coronary angiography and the role of beta-blocker therapy; To describe the clinical and anatomical characteristics of patients presenting with MB; To determine the impact of cardiovascular medications on symptoms in patients with MB; To describe the anatomical and clinical features associated with the invasive evidence of ischemia in patients with MB; To assess the relation between invasively documented ischemia and clinical manifestations in patients with the MB. Inclusion Criteria: patients referred to undergo ICA (for both elective or urgent indications) for suspected coronary artery disease found to have an MB with or without other epicardial lesions amenable to revascularization; Age above 18 y.o.; Ability to provide Informed Consent. Exclusion Criteria are Patients with life expectancy below 12 months and Patients with severe valvular heart disease. The primary endpoint is the incidence of MACE defined as the composite of cardiac death, myocardial infarction, cardiac hospitalization, and target vessel revascularization. The secondary endpoint is evaluating the Rate of patients with SAQ < 70 and the Rate of patients with "high-risk features" on CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to undergo ICA (for both elective or urgent indications) for suspected coronary artery disease found to have a myocardial bridge with or without other epicardial lesions amenable to revascularization
* Age above 18 y.o.
* Ability to provide Informed Consent

Exclusion Criteria:

* Patients with life expectancy below 12 months
* Patients with severe valvular heart disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with suspected coronary artery disease found to have a myocardial bridge with or without other epicardial lesions amenable to revascularization
Sampling Method: Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2022-03-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
Incidence of MACE | 2 years follow up
  Incidence of MACE defined as the composite of cardiac death, myocardial infarction, cardiac hospitalization and target vessel revascularization

SECONDARY OUTCOMES:
Rate of patients with SAQ < 70 | 2 years follow up
Rate of patients with "high risk features" on CT scan | 2 years follow up
  High risk features

CONTACTS AND LOCATIONS:
Locations (5):
- Italy (5):
  - Arcispedale S. Anna, Azienda Ospedaliero - Universitaria di Ferrara, Ferrara, Italia
  - Policlinico S. Martino IRCCS, Università di Genova, Genova, Italia
  - Centro Cardiologico Monzino IRCCS, Milan, Italia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, Italia
  - Policlinico Universitario Tor Vergata Fondazione PTV, Roma

IPD SHARING:
Plan to Share IPD: Undecided